CLINICAL TRIAL: NCT03406039
Title: Testing the Efficacy of an Online Self-Help Treatment for Comorbid Alcohol Misuse and Emotional Problems in Young Adult Canadians: A Randomized Controlled Trial (RCT)
Brief Title: Testing the Efficacy of an Online Integrated Treatment for Comorbid Alcohol Misuse and Emotional Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2017:128
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Emotional Disorder; Cognitive Behavioural Therapy; Motivational Interviewing; Online Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: A two-arm RCT will be conducted to evaluate the proposed online intervention. Eligible participants will be randomized to either the online integrated treatment condition, or the psycho-educaton (i.e., control) condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Online CBT and MI (Experimental): Participants in this arm will be given access to the online integrated treatment.
  Interventions: Behavioral: Integrated Online CBT and MI
- Psychoeducation (Control) (No Intervention): The control group will be provided with psychoeducational resources about alcohol and mental illness.

INTERVENTIONS:
Behavioral: Integrated Online CBT and MI — The treatment condition will have access to 12 treatment modules and have 8-weeks to complete them. The content of all modules is derived from Cognitive Behavioural Therapy and Motivational Interviewing. Through module engagement, young adults will identify goals related to alcohol use and mood, learn strategies to cope with alcohol cravings, triggers, and social pressures, and learn how to prevent relapse. There will also be several modules to target anxiety and depression, focusing on strategies designed to help reduce negative thinking and worry, increase behavioural activation, and increase self-care (e.g., sleep hygiene).Participants will have immediate access to all modules, and it will be recommended that they work through the modules sequentially.
  Arms: Integrated Online CBT and MI

SUMMARY:
Considering the high comorbidity between alcohol use disorders and emotional problems, there is currently a need for accessible, integrated treatments designed to target both disorders simultaneously. Evidence suggests that the combined use of Cognitive Behavioural Therapy (CBT) and Motivational Interviewing (MI) may be effective at reducing the combined symptoms of the two disorders. However, much of the empirical work has focused on testing the usefulness of CBT/MI for alcohol misuse and comorbid depression, and the majority of these studies involve in-person treatment. Therefore, additional empirical research is required to determine the efficacy of combined CBT and MI for alcohol use and both anxiety and depression using an online intervention. This may help inform future treatments in this domain, and potentially be able to inform the development of online, accessible interventions for this population.

Participants (N = 214) with elevated levels of alcohol use and emotional problems will be recruited from Central and Eastern Canada. Participants will be randomly assigned to either the treatment group (i.e., combined CBT and MI), or the psycho-educational control group. Individuals in the treatment group will be given 8-weeks to work through 12 online modules. Throughout the modules, participants will identify goals related to alcohol use and mood, learn strategies to cope with alcohol cravings, triggers, and social pressures, and learn how to prevent relapse. Modules will also include content designed to target anxiety and depression, focusing on strategies designed to help reduce negative thinking and worry, increase behavioural activation, and increase self-care (e.g., relaxation techniques, sleep hygiene). Participants randomly assigned to the control (i.e., psycho-education) condition will receive links to websites that provide general psychoeducation about alcohol and mental illness. All participants will complete online assessment measures at baseline, at the end of treatment, and at follow-up approximately 4 months later) in order to assess the efficacy of the treatment. At the end of the study, individuals in the control group will be given full access to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18 and 35 years old
* Reporting at least moderate difficulties with alcohol indicated by a score >3 (for women) and <4 (for men) on the first three items of the Alcohol Use Disorders Identification Test [AUDIT], known as the AUDIT-C
* Reporting at least moderate depression and/or anxiety symptoms indicated by a score >16 on the Center for Epidemiological Studies Depression Scale [CES-D] and/or a score of >5 on the Generalized Anxiety Disorder Scale-7 [GAD-7]
* Fluency in English
* Have weekly Internet access

Exclusion Criteria:

* Self-reported engagement in other psychological or pharmacological treatments for alcohol misuse and/or depression/anxiety (with the exception of stable anti-depressants)
* Elevated suicidality (defined as scoring greater than "minimal risk" on a screener)
* Current psychosis or mania

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 273 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Change in Alcohol Use | Participants will be assessed using the TLFB at three time points: at baseline (i.e., prior to treatment; T0), immediately following the 8-week treatment (T1), and at follow-up (i.e., 24 weeks from baseline, 16 weeks from end of treatment, T2).
  Timeline Follow-Back (TLFB; Sobell & Sobell, 1992) - designed to assess the number of standard drinks consumed during a 30-day period. Participants will be asked to report on the number of drinks consumed daily in the form of a calendar. The TLFB has been shown to provide reliable and valid estimates of alcohol use, and is widely used in basic and treatment studies.

SECONDARY OUTCOMES:
Depression | Levels of depression will be assessed at all three time points. T0 - baseline (i.e., 0 days, 0 weeks, 0 months), T1 - end of treatment (i.e., 8 weeks), and T2 - follow up (i.e., 16 weeks from end of treatment).
  Center for Epidemiological Studies Depression Scale (CES-D; Radloff, 1977), a 20-item self-report questionnaire used to indicate depression severity.
Anxiety | Levels of anxiety will be assessed at all three time points. T0 - baseline (i.e., 0 days, 0 weeks, 0 months), T1 - end of treatment (i.e., 8 weeks), and T2 - follow up (i.e., 16 weeks from end of treatment).
  Generalized Anxiety Disorder Scale-7 (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006), a 7-item self-report questionnaire used to measure the severity of anxiety symptoms.
Clinically Significant and Combined Reduction of Alcohol Use and Comorbid Emotional Problems | Combined changes will be assessed at all three time points. T0 - baseline (i.e., 0 days, 0 weeks, 0 months), T1 - end of treatment (i.e., 8 weeks), and T2 - follow up (i.e., 16 weeks from end of treatment).
  We will also use a combined outcome to look clinically significant reductions in alcohol misuse and depression or anxiety. Specifically, a short version of the Alcohol Use Disorders Identification Test (AUDIT; Saunders et al., 1993, referred to as AUDIT-C) will be used, where falling below 4 for women and 5 for men would reflect that participants are no longer drinking hazardously. Similarly, falling below 16 on the CES-D OR 5 on the GAD-7 would reflect that participants are no longer experiencing moderate emotional symptoms. A binary outcome will be created for participants scoring below the AUDIT-C cut-off AND the cut-off for either depression OR anxiety (coded as 1) versus those scoring above cut-offs (coded as 0).
Quality of Life | Quality of life will be assessed at all three time points. T0 - baseline (i.e., 0 days, 0 weeks, 0 months), T1 - end of treatment (i.e., 8 weeks), and T2 - follow up (i.e., 16 weeks from end of treatment).
  World Health Organization Quality of Life assessment (WHOQOL-BREF; The WHOQOL Group, 1998), a 26-item self-report measure that assesses functionality in various life domains (i.e., physical and psychological health, social relationships, environment). A sum score will be used to assess overall quality of life at all assessments (T0-T2).
Drug Use | Drug use will be assessed at all three time points. T0 - baseline (i.e., 0 days, 0 weeks, 0 months), T1 - end of treatment (i.e., 8 weeks), and T2 - follow up (i.e., 16 weeks from end of treatment).
  Participants' use of other drugs in addition to alcohol will also be included as outset continuous moderators and will be assessed using the National Institute on Drug Abuse Alcohol, Smoking, and Substance Involvement Screening Test (NIDA ASSIST; National Institute on Drug Abuse, 2009). Examples of these additional substances include cannabis, cocaine, prescription medication, methamphetamine, and opioids.
Motivation | Motivation will be assessed at all three time points. T0 - baseline (i.e., 0 days, 0 weeks, 0 months), T1 - end of treatment (i.e., 8 weeks), and T2 - follow up (i.e., 16 weeks from end of treatment).
  Participants' level of motivation will be assessed at all assessment points. Motivation for change will be assessed along three dimensions: importance, confidence, and readiness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frohlich JR, Rapinda KK, Schaub MP, Wenger A, Baumgartner C, Johnson EA, O'Connor RM, Vincent N, Blankers M, Ebert DD, Hadjistavropoulos H, Mackenzie CS, Keough MT. Efficacy of an Online Self-Help Treatment for Comorbid Alcohol Misuse and Emotional Problems in Young Adults: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Nov 1;7(11):e11298. doi: 10.2196/11298. PMID 30389649

DOCUMENTS (3):
  • Study Protocol (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT03406039/Prot_003.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT03406039/SAP_004.pdf
  • Informed Consent Form (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT03406039/ICF_005.pdf